CLINICAL TRIAL: NCT03688490
Title: Aquagenic Pruritus Among Patients With Myeloproliferative Syndromes (in English) Prurit Aquagénique Dans Les SYndromes MyéloProLifEratifs (in French)
Brief Title: Clinical Characteristics of Aquagenic Pruritus in Patients With Myeloproliferative Neoplasms
Acronym: PASYMPLE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PASYMPLE
Record Dates: First submitted 2018-09-20; First posted 2018-09-28 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2018-08

CONDITIONS: Myeloproliferative Disorder
Keywords: aquagenic pruritus
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Description of the characteristics of aquagenic pruritus expressed by patients suffering from myeloproliferative neoplasms.

Prospective work based on the distribution of a dedicated questionnaire.

DETAILED DESCRIPTION:
Patients with myeloproliferative neoplasms identified and followed in our Institution (Brest University Hospital). Patients could be followed for polycythemia vera or essential thrombocythemia or myelofibrosis.

Distribution of the questionnaire to each patients with myeloproliferative neoplasms (treated or not) suffering from aquagenic pruritus.

Analyse of each characteristic of the aquagenic pruritus by a statistician and publication at the end.

ELIGIBILITY:
Inclusion Criteria:

* patients followed with myeloproliferative neoplasms
* suffering from aquagenic pruritus

Exclusion Criteria:

* Unable to fulfil the questionnaire
* No written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed for myeloproliferative neoplasms in our Institution (Brest University Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-07-17 (Actual); Primary Completion 2013-11-04 (Actual); Study Completion 2013-11-04 (Actual)

PRIMARY OUTCOMES:
Intensity of the pruritus | 15 days
  Analogic Visual Scale, from 0 to 10, Worse if >6

SECONDARY OUTCOMES:
Duration of the pruritus | 15 days
  Timing expresses in minutes

CONTACTS AND LOCATIONS:
Overall Officials: IANOTTO Jean-Christophe, MD, PhD, Principal Investigator — Hématologie Clinique-Institut de Cancéro-Hématologie

REFERENCES:
- [Result] Le Gall-Ianotto C, Brenaut E, Gouillou M, Lacut K, Nowak E, Tempescul A, Berthou C, Ugo V, Carre JL, Misery L, Ianotto JC. Clinical characteristics of aquagenic pruritus in patients with myeloproliferative neoplasms. Br J Dermatol. 2017 Jan;176(1):255-258. doi: 10.1111/bjd.14809. Epub 2016 Dec 22. No abstract available. PMID 27291777